CLINICAL TRIAL: NCT05046691
Title: Mindfulness, Compassion and Self-compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Shui-fong, Director, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHongKong (PandA)
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Issue
Keywords: mindfulness; teacher mental health; compassion; self-compassion; common humanity; mindfulness-based intervention for teachers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 8-week .b Foundations course
  Interventions: Behavioral: 8-week mindfulness program
- Wait-list control (No Intervention): Participants in wait-list control group will receive the same intervention, two months after their counterparts in experimental group completed the intervention.

INTERVENTIONS:
Behavioral: 8-week mindfulness program — The .b Foundations course is an 8-week mindfulness program developed by Mindfulness in Schools Project (MiSP) for school teachers and personnel. It includes a taster session and 8 weekly sessions. Each session lasts for 1.5 hours with a specific theme (e.g. Lesson 1 waking up from autopilot). Formal and informal mindfulness practices (e.g. mindful eating, body scan, mindful walking, habit releaser etc.), psychoeducation, cognitive exercises, inquiry, and home practice are involved.
  Arms: Intervention group

SUMMARY:
Teachers in Hong Kong are susceptible to professional stress and its associated psychosomatic illnesses. To enhance teachers' well-being, mindfulness training is conducted in local schools. The present study is a randomized controlled trial to explore 1) the relationship between mindfulness, common humanity, self-compassion, compassion, and well-being of school teachers; 2) whether mindfulness and common humanity are the antecedents of self-compassion and compassion; 3) the conditions under which compassion and self-compassion are highly correlated. Participants will be randomized to either intervention (8-week .b Foundations course) or waiting-list control condition. They will complete an online survey before (baseline), after (post-intervention), and two-months (follow-up) after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or above
* Working in local schools or education institutions
* Willing to participate in mindfulness training voluntarily

Exclusion Criteria:

* Experiencing severe or unstable mental health condition currently
* Completed 8-week mindfulness training previously
* Unwilling to go by random assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in General Health | Baseline, Immediately after intervention, Two-months after intervention
  General Health Questionnaire (GHQ), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Stress | Baseline, Immediately after intervention, Two-months after intervention
  Perceived Stress Scale (PSS), 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)

SECONDARY OUTCOMES:
Change in Positive affect | Baseline, Immediately after intervention, Two-months after intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Negative affect | Baseline, Immediately after intervention, Two-months after intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Compassion | Baseline, Immediately after intervention, Two-months after intervention
  Compassion scale, 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Self-compassion | Baseline, Immediately after intervention, Two-months after intervention
  Self-compassion scale, 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Common humanity | Baseline, Immediately after intervention, Two-months after intervention
  Common Humanity scale, 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Mindfulness | Baseline, Immediately after intervention, Two-months after intervention
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey Club "Peace and Awareness" Mindfulness Culture in Schools Initiative, Faculty of Social Sciences, The University of Hong Kong, Hong Kong, Hong Kong